CLINICAL TRIAL: NCT05518526
Title: Phase 1b/2 Study of Liposomal Annamycin (L-Annamycin) in Subjects With Previously Treated Soft-Tissue Sarcomas (STS) With Pulmonary Metastases (ANNA-SARC)
Brief Title: Phase 1b/2 Study of Liposomal Annamycin (L-Annamycin) in Subjects With Previously Treated Soft-Tissue Sarcomas (STS) With Pulmonary Metastases
Acronym: ANNA-SARC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIO-0002
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Soft Tissue Sarcoma; Pulmonary Metastasis
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- L-Annamycin (Experimental)
  Interventions: Drug: Liposomal Annamycin (L-Annamycin)

INTERVENTIONS:
Drug: Liposomal Annamycin (L-Annamycin) — Study drug consists of L-Annamycin as a lyophilised powder in 50-mL single-use vials containing 45 mg of L-Annamycin must be reconstituted with 45 mL of 0.9% sodium chloride injection between 34 to 42℃, USP, and then diluted 1:1 with 0.9% sodium chloride injection between 34 to 42℃ in non-polyvinyl chloride IV bags before intravenous infusion. The dose of L-Annamycin will be intravenously applied during 2 hours infusion on D1, D8, and D15 of each 28-day cycle (up to Cycle 6th).

SUMMARY:
This study is a multi-centre, open-label, single-arm, 3+3 Phase 1b/ and Phase II. Phase 1b is aimed to determine the maximum-tolerated dose (MTD)/Recommended Phase 2 Dose (RP2D) based on safety reporting. The RP2D is a multifactorial endpoint that considers toxicity as well as additional determinants (e.g. efficacy, pharmacodynamics) to define the optimal Phase 2 dose. Phase 2 will explore the efficacy of L-Annamycin at RP2D for treating soft tissue sarcomas (STS) subjects with lung metastases, for which chemotherapy is considered appropriate.

DETAILED DESCRIPTION:
The project aims to conduct a Phase 1b/2 clinical trial using liposomal Annamycin (L-Annamycin) in subjects diagnosed with soft tissue sarcoma (STS) in the stage of unresectable pulmonary dissemination after the failure of at least one line of prior systemic treatment.

The most common localisation of metastatic lesions in STS is the lungs (refer to this as a "sanctuary site" for STS). Furthermore, although the most common dosing regimen for other anthracyclines (typically, doxorubicin) in the treatment of STS has historically been once every three weeks, preclinical testing of L-Annamycin suggests that weekly dosing of L-Annamycin may be more beneficial, as well as it seems to be both safer and more effective than alternative schedules.

Therefore, this Phase Ib/II clinical trial will test the hypothesis that L-Annamycin administration in monotherapy in the weekly schedule (D1, D8, D15 in 28-day cycles) is safe and has the pharmacodynamic (PD) potential to restore and enhance tumour responses in anthracycline-pre-treated subjects with advanced and/or metastatic STS until disease progression, unacceptable toxicities, or subject consent withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is ≥18 years old at the time of signing informed consent.
2. The subject has an ECOG performance status ≤2 with an estimated life expectancy of greater than three months.
3. The subject has a pathologically confirmed diagnosis of STS (including the following pathological subtypes: liposarcoma, leiomyosarcoma, synovial sarcoma, angiosarcoma, undifferentiated pleomorphic sarcoma, myxofibrosarcoma, malignant peripheral nerve sheath tumour, malignant solitary fibrous tumour, and pleomorphic RMS), and documented lung metastases that are considered eligible for chemotherapy and not eligible for potentially curative surgical resection.
4. The subject must have measurable disease in the lung, defined as, at a minimum, one lesion that can be accurately measured in at least one dimension of >10 mm. Subjects with the extra-pulmonary disease are eligible.
5. The subject had prior anthracycline therapy (cumulative dose of ≤450 mg/m2) for their disease and has shown the progression of the disease before study entry - for phase II trial maximum of three previous lines of therapy (adjuvant/neoadjuvant regimen is counted as one line of systemic treatment)
6. At least two weeks must have passed following treatment for their disease with chemotherapy, investigational therapy, targeted agents, biological agents, immune modulators, and any toxicities must have resolved to ≤ grade 1 or previous baseline levels no more than four weeks after completing therapy (except alopecia and polyneuropathy).
7. The subject must have adequate laboratory results, including the following:

   1. Absolute neutrophil count ≥ 1500/mL and platelets ≥100,000/mL
   2. Hemoglobin ≥8.0 g/dL
   3. Adequate renal function (The Cockcroft-Gault equation will be used to estimate creatinine clearance. This equation is as follows: Creatinine clearance in milliliters per minute= [140-age] x body weight [kg]/72 x plasma creatinine [mg/dL]; multiplied by 0.85 for women. By using this equation, adequate renal function will be deemed to be a creatinine clearance of greater than 60 mL/minute)
   4. Bilirubin ≤1.5 x ULN (unless due to Gilbert's syndrome)
   5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5 x ULN in subjects with liver metastases)
8. The subject is able to understand and sign the informed consent document, can communicate with the Investigator, and can understand and comply with the requirements of the protocol.
9. Vaccinated with a live vaccine within 28 days prior to the first dose of the study drug. COVID-19 vaccination with mRNA or replication incompetent viral vector vaccines and annual inactivated influenza vaccines are permitted.
10. All subjects (men and women) agree to practise effective contraception during the entire study period and after discontinuing the study drug unless documentation of infertility exists.

    1. Sexually active, fertile women must use two effective forms of contraception (abstinence, intrauterine device, oral contraceptive, or double barrier device) from the time of informed consent and until at least six months after discontinuing the study drug.
    2. Sexually active men and their sexual partners must use effective contraceptive methods from the time of informed consent until at least six months after discontinuing the study drug.

Exclusion Criteria:

1. The subject has any condition that, in the opinion of the Investigator, places the subject at unacceptable risk if they were to participate in the study.
2. Metastases to the central nervous system
3. The subject has left ventricular ejection fraction (LVEF) <50%, valvular heart disease, or severe hypertension not controlled by medical therapy. Cardiac subjects with a New York Heart Association classification of 3 or 4 will be excluded, as will those with recent (≤ 6 months) myocardial infarction, unstable angina, or symptomatic congestive heart failure. The subject has a baseline QT/QTc interval >480 msec, a history of additional risk factors for torsade des pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome) and use of concomitant medications that significantly prolong the QT/QTc interval.
4. The subject has clinically relevant serious comorbid medical conditions including, but not limited to active infection, known positive status for human immunodeficiency virus and/or active hepatitis B or C, cirrhosis, or psychiatric illness/social situations that would limit compliance with study requirements.
5. The subject is pregnant, lactating, or not using adequate contraception.
6. The subject has a known allergy to study drug or excipients.
7. The subject is required to use moderate or strong inhibitors and inducers of cytochrome P450 (CYP) family enzymes CYP3A and CYP2B and transporters that cannot be held three days before treatment and on the day of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Recommended Phase 2 Dose (RP2D). | up to 24 weeks
Phase II: 3-month Progression-Free Survival (PFS). | 3 months

SECONDARY OUTCOMES:
Phase Ib/II: Overall response rate (ORR): complete response (CR) and partial response (PR) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw, Mazovian, Poland